CLINICAL TRIAL: NCT06587698
Title: Sitagliptin or BeiDouGen Capsule Improve the Pregnancy Outcome in Patients with PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2024342
Record Dates: First submitted 2024-07-25; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Sitagliptin Phosphate; xin-kang

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sitagliptin (Other): 100mg/day Sitagliptin by oral for 3 months
  detail：1 piece(100mg) at morning
  Interventions: Drug: Sitagliptin
- BeiDouGen (Other): 120mg/day BeiDouGen capsule by oral for 3 months
  detail：2 piece(30mg) at morning and night
  Interventions: Drug: BeiDouGen
- Sitagliptin+BeiDouGen (Other): 100mg/day Sitagliptin+120mg/day BeiDouGen capsule by oral for 3 months
  detail：1 piece(100mg) Sitagliptin and 2 piece(30mg) BeiDouGen capsule at morning 2 piece(30mg) BeiDouGen capsule at night
  Interventions: Drug: Sitagliptin+BeiDouGen

INTERVENTIONS:
Drug: Sitagliptin — 100 mg QD for 3 month
  Other Names: brand name:Jie Nuo Wei
  Arms: Sitagliptin
Drug: BeiDouGen — 60 mg BID for 3 month
  Other Names: brand name:Kang xin
  Arms: BeiDouGen
Drug: Sitagliptin+BeiDouGen — 100 mg Sitagliptin QD plus BeiDouGen 60 mg BID for 3 month
  Other Names: brand name:Jie Nuo Wei and Kang xin
  Arms: Sitagliptin+BeiDouGen

SUMMARY:
This study will be carried out under the guidance of professional doctor, patients with PCOS will be treated with Sitagliptin or BeiDouGen capsule or both two to assess their ovarian function and reproductive outcomes, and compare the effect of different treatment methods, which will provide the basis for PCOS intervention strategy and related research

DETAILED DESCRIPTION:
Subject Recruitment and Grouping This study adopts an open-label randomized controlled trial design. We plan to recruit a total of 300 patients with polycystic ovary syndrome (PCOS) by introducing the purpose, benefits, and risks of the study to patients in medical or examination units. PCOS patients who meet the inclusion criteria and do not meet the exclusion criteria will be registered and given a questionnaire by the research staff after signing the informed consent form. Physical and blood examinations will be conducted, and electronic randomization will be performed using the Redcap platform.

Intervention Measures After signing the informed consent form, enrolled patients will be randomly assigned to the Sitagliptin intervention group, the Bei Dou Gen intervention group, or the combination therapy group of Sitagliptin and Bei Dou Gen. Before enrollment, all three groups will undergo baseline assessments including blood routine, liver and kidney function, blood lipids, endocrine hormones, gynecological ultrasound, liver ultrasound, and physical examinations.

For participants in the Sitagliptin intervention group, Sitagliptin will be administered orally at a dose of 100 mg once daily for a treatment period of three months. Participants in the Bei Dou Gen intervention group will receive Bei Dou Gen capsules orally at a dose of 60 mg twice daily for a treatment period of three months. Participants in the combination therapy group will receive both Sitagliptin at a dose of 100 mg once daily and Bei Dou Gen capsules at a dose of 60 mg twice daily for a treatment period of three months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20-40 years who plan to conceive or are infertile in our center.

Diagnosed with PCOS according to the Rotterdam criteria: Diagnosis of PCOS can be made if two out of the following three criteria are met: (1) Oligoovulation or anovulation, (2) Clinical or biochemical signs of hyperandrogenism, (3) Polycystic ovaries on ultrasound examination.

Patients who are regularly followed up at our clinic. No participation in other research projects currently or in the past 3 months.

Exclusion Criteria:

Exclusion criteria (any of the following criteria met will result in exclusion):

Pregnant, lactating, or postmenopausal women. Taking weight loss medications or undergoing weight loss surgery in the past 3 months or currently.

Food allergies. Other diseases that may cause hyperandrogenism or ovulation abnormalities (e.g., Cushing's syndrome, non-classical congenital adrenal hyperplasia, tumors secreting androgens in the ovaries or adrenal glands, functional hypothalamic amenorrhea, thyroid diseases, hyperprolactinemia, premature ovarian insufficiency, etc.).

Use of insulin, hypoglycemic drugs, or beta-blockers in the past 3 months. Patients with chronic diseases such as hypertension, gout, hyperuricemia, diabetes, etc., requiring regular medication.

Use of glucocorticoids, anti-androgenic drugs, oral contraceptives, ovulation-inducing drugs, weight loss drugs, or other medications affecting hormone levels, appetite, and carbohydrate metabolism in the past 2 months.

Patients with liver cirrhosis or various severe liver diseases (alanine aminotransferase and/or aspartate aminotransferase exceeding 3 times the upper limit of normal), patients with abnormal renal function (serum creatinine exceeding the upper limit of normal), patients with kidney disease or other diseases requiring control of protein intake.

Patients currently or previously with severe cardiovascular and cerebrovascular diseases that may interfere with the normal conduct of the trial (such as heart failure, myocardial infarction, cerebral infarction, acute myocarditis, severe arrhythmias, patients undergoing interventional therapy, etc.).

Patients currently with severe gastrointestinal diseases such as gastrointestinal ulcer bleeding, chronic diarrhea, or who have undergone gastrointestinal resection surgery, which may affect nutrient absorption.

Patients with infectious diseases such as hepatitis B e antigen-positive, active pulmonary tuberculosis, or HIV.

Cancer patients or those who have received radiation and chemotherapy within the past five years.

Patients with any psychological or psychiatric disorders requiring medication, including epilepsy patients or those undergoing antiepileptic treatment, patients using antidepressants, etc.

Daily alcohol consumption exceeding 15g. Smoking habit

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | through study completion, an average of 2 year
  the pregnancy situation among volunteers

SECONDARY OUTCOMES:
DHEA | before and after intervention（3 month）
  dehydroepiandrosteron in serum during menstruation period
total testosterone | before and after intervention（3 month）
  total testosterone in serum during menstruation period
FAI | before and after intervention（3 month）
  Free testosterone index calculated by total testosterone and SHBG
LH/FSH | before and after intervention（3 month）
  the rate between LH and FSH
ovarian volume | before and after intervention（3 month）
  the size is measured by ultrasound
number of antral follicles | before and after intervention（3 month）
  the number is is measured by ultrasound during menstruation period
Number of retrieved eggs | after intervention（3 month）
  the number is observed during the surgery
number of mature eggs (MII) | after intervention（3 month）
  observed the state of oocytes during the IVF laboratory
fertilization rate | after intervention（3 month）
  observed the state of oocytes during the IVF laboratory
number of usable embryos, | after intervention（3 month）
  observed the state of embryos during the IVF laboratory
number of high-quality embryos | after intervention（3 month）
  observed the state of embryos during the IVF laboratory
GLP-1 levels | before and after intervention（3 month）
  measure it in the serum
fasting glucose | before and after intervention（3 month）
  measured by glucometer
OGTT | before and after intervention（3 month）
  measured by glucometer
HOMA index | before and after intervention（3 month）
  calculated by glucose and INS

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Study Chair — the third hospital of peking universry
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No